CLINICAL TRIAL: NCT02574338
Title: Cervical Ripening: A Comparison Between Intravaginal Misoprostol Tablet and Intracervical Foley's Catheter and Subsequent Induction of Labor, Safety and Efficacy in Federal Teaching Hospital Abakaliki, Ebonyi State, Nigeria.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nwali Matthew Igwe (Other Government)
Responsible Party: Sponsor-Investigator, Nwali Matthew Igwe, Dr, Federal Teaching Hospital Abakaliki
Organization: Federal Teaching Hospital Abakaliki (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSFC-2015-CT
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Cervical Ripening and Induction of Labor
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group - 1 Foley's Catheter (Active Comparator): will have cervical ripening with intracervical extraamniotic Foley's catheter for 24 hours
  Interventions: Device: Foley's Catheter
- Group - 2 Prostaglandin E1 Analogue (Active Comparator): will have cervical ripening with intravaginal misoprostol inserted into the posterior fornix every six hours to a maximum of four doses (24 hours)
  Interventions: Drug: prostaglandin E1 analogue

INTERVENTIONS:
Device: Foley's Catheter — intracervical extraamniotic Foley's catheter
  Arms: group - 1 Foley's Catheter
Drug: prostaglandin E1 analogue — intravaginal misoprostol
  Other Names: Misoprostol
  Arms: Group - 2 Prostaglandin E1 Analogue

SUMMARY:
The aim of this study is to compare the effectiveness and safety of Foley's catheter and misoprostol in cervical ripening.

DETAILED DESCRIPTION:
This is a randomized clinical study which will be made up of two arms or groups. The first arm or group - 1 will have cervical ripening with intracervical extraamniotic Foley's catheter while group - 2 will have cervical ripening with intravaginal misoprostol. The parturients will be randomly selected by simple lottery and recruited into the two arms of the study. Each parturient will pick by simple lucky dip from a pool of folded papers with inscription group 1 or group 2 in a bag in a double blinded manner and will be recruited into the group picked among the two arms of the study. The Bishop's score of the cervix will be accurately determined and documented before cervical ripening. Bishop's score of ≥6 will be considered ripe. Oxytocin will be used for induction or augmentation of labor as required.

ELIGIBILITY:
Inclusion Criteria:

* Parturients who gave consent
* has low bishop score (≤5)
* term singleton cephalic presenting fetus
* intact membranes
* no contraindication to vaginal delivery

Exclusion Criteria:

* those who refused consent
* preterm delivery
* vaginal infection
* non-cephalic presentation
* multiple gestation
* low lying placenta/previa,
* vaginal bleeding,
* previous cesarean section
* rupture of membranes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Bishop Score of 6 or more | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Teaching Hospital, Abakaliki, Abakaliki, Ebonyi State, Nigeria

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264